CLINICAL TRIAL: NCT01964846
Title: The Effect of Resveratrol and Curcumin on Postprandial Inflammation in Men and Postmenopausal Women
Brief Title: Effect of Antioxidant Intake on Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Atrium Innovations (Industry)
Responsible Party: Principal Investigator, Charles Couillard, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: INAF-2013-023
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Effect of Resveratrol and Curcumin on Inflammation
Keywords: inflammation; high fat meal; resveratrol; curcumin; gene expression
MeSH Terms: conditions — Inflammation | interventions — Resveratrol; Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol, curcumin (Experimental): Subjects will take 2 capsules of resveratrol and curcumin. Thirty (30) minutes later, subjects will be given an oral lipid tolerance test in the form of a fat-rich meal. Blood samples will be collected at different time points.
  Interventions: Dietary Supplement: Resveratrol, curcumin
- Placebo (Placebo Comparator): Subjects will take 2 capsules of Placebo. Thirty (30) minutes later, subjects will be given an oral lipid tolerance test in the form of a fat-rich meal. Blood samples will be collected at different time points.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol, curcumin
  Arms: Resveratrol, curcumin
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The general objective of this project is to investigate the acute effect of consuming a dietary supplement combining resveratrol and curcumin on the inflammatory response following the consumption of a high-fat meal in healthy subjects with slightly elevated waist circumference.

The study will be undertaken according to a double-blind, cross over, randomized, placebo controlled design and will be conducted at the Institute of Nutrition and Functional Foods (INAF) of Laval University. The study will involve a total of 20 healthy subjects (10 men and 10 women. Included subjects will undergo an 6-hour oral fat tolerance, on two separate occasions (one time following dietary supplement consumption and one time following consumption of a placebo). The two test days will be separated by maximum of two weeks. The outcomes are the changes in the plasma levels of inflammatory cytokines in their gene expression.

DETAILED DESCRIPTION:
There is increasing evidence showing that inflammation is implicated in the pathogenesis of numerous chronic conditions and cardiovascular disease (CVD). Also, high-fat meals have been shown to induce postprandial oxidative stress and inflammation. Polyphenols are compounds found ubiquitously in plants and are known to regulate many processes like plant growth, reproduction, seed germination as well as resistance to pathogens and predators. They are present in fruits and vegetables and exhibit favorable physiological effects that even if they remain not fully understood, still allow the classification of phenolic compounds as antiinflammatory molecules.

Resveratrol is a polyphenol that is found in berries, grapes and red wine among others. Interest for resveratrol as a health-promoting molecule has flourished in recent years as it has been shown to prevent co-morbidities associated with diabetes and CVD. Evidence of the physiological benefits of resveratrol in humans is somewhat limited, but nonetheless supports an antiinflammatory action.

There is also an increasing body of evidence supporting the role of curcumin, a polyphenol from the curcuminoid family, as a modulator of the inflammatory pathway.These observations underline the anti-inflammatory potential of curcumin and how it may serve in the prevention and treatment of chronic conditions like diabetes and CVD.

The general objective of this project is to investigate the acute effect of consuming dietary supplement combining resveratrol and curcumin on the inflammatory response following the consumption of a high-fat meal in healthy individuals with slightly elevated waist girth.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women aged between 45-70 years
* When applicable, menopause will be defined as the absence of menses for at least 1 year
* Weight stable (for at least three (3) months)
* Otherwise healthy individuals
* No medication
* Waist circumference >=94 cm for men or >=80 cm for women
* With one (and no more than one) of the following:
* triglycerides >=1.7 mmol/L
* HDL-c <=1.03 mmol/L for men and <=1.29 mmol/L for women
* fasting glucose >=5.6 mmol/L
* systolic blood pressure >=130 or diastolic blood pressure >=85 mmHg

Exclusion Criteria:

* Diagnosis of hypertension, CVD, T2D or endocrine disorders
* Aversion/intolerance to spice
* ≥ 3 risk factors for the metabolic syndrome (IDF)
* Fasting triglycerides > 4 mmol/L

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in blood levels of anti- and pro-inflammatory markers | At the end of the two lipid tolerance tests [week0; week 2]

SECONDARY OUTCOMES:
Change in the expression of anti- and pro-inflammatory genes in total blood RNA from white blood cells (WBC) | At the end of the two lipid tolerance tests [week0; week 2]

CONTACTS AND LOCATIONS:
Overall Officials: Charles Couillard, PhD, Principal Investigator — INAF - Université Laval
Locations (1):
- Institute on Nutrition and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Vors C, Couillard C, Paradis ME, Gigleux I, Marin J, Vohl MC, Couture P, Lamarche B. Supplementation with Resveratrol and Curcumin Does Not Affect the Inflammatory Response to a High-Fat Meal in Older Adults with Abdominal Obesity: A Randomized, Placebo-Controlled Crossover Trial. J Nutr. 2018 Mar 1;148(3):379-388. doi: 10.1093/jn/nxx072. PMID 29546309